CLINICAL TRIAL: NCT07010939
Title: A Prospective Multi-modal Cohort Study of Local Treatment-related Toxicities and Quality of Life in Chinese Breast Cancer Patients (PERSEVERE)
Brief Title: A Study of Treatment-Related Toxicities and Quality of Life After Local Therapy in Chinese Breast Cancer Patients
Acronym: PERSEVERE
Status: Recruiting | Type: Observational
Sponsor: FangYi (Other)
Responsible Party: Sponsor-Investigator, FangYi, Chief Physician and Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: 245194799
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms; Quality of Life (QOL); Toxicities; Breast Diseases
Keywords: Breast Neoplasms; Treatment-Related Toxicities; Quality of Life; Patient-Reported Outcomes; Prospective Study
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral blood: Plasma and peripheral blood mononuclear cells (PBMCs) will be collected using EDTA anticoagulant tubes. Plasma will be processed and stored at -80°C for future biomarker and multi-omics analyses. PBMCs will be isolated and cryopreserved in liquid nitrogen.
  Tumor tissue: Formalin-fixed and/or fresh-frozen samples of tumor tissue will be collected during breast cancer surgery.
  Adjacent normal breast tissue: When available, paired peritumoral normal tissue samples will also be collected during surgery.
  All samples will be stored in a centralized biobank under standard quality-controlled conditions for future translational research related to treatment-related toxicities and recovery in breast cancer patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early-Stage Breast Cancer Patients Receiving Local Therapy: This group includes people diagnosed with stage I to III breast cancer who are receiving local therapy with curative intent. Local therapy in this study includes surgery, as well as systemic treatments given before or after surgery, such as:
  Neoadjuvant therapy (for example, chemotherapy or targeted therapy given before surgery)
  Adjuvant therapy (for example, chemotherapy, radiotherapy, endocrine therapy, or targeted therapy given after surgery)
  This is an observational study. There is no experimental intervention. All participants will undergo baseline assessments, including clinical evaluations, laboratory tests, patient-reported outcome questionnaires, and biospecimen collection. Participants will then be followed over time to monitor treatment-related toxicities and changes in quality of life.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — At baseline, participants will undergo peripheral blood collection using EDTA tubes. A total of 10 mL of venous blood will be collected and processed into plasma and peripheral blood mononuclear cells (PBMCs). Plasma samples will be stored at -80°C, and PBMCs will be cryopreserved in liquid nitrogen. These samples will be used for future biomarker discovery, multi-omics analysis, and studies of biological mechanisms underlying treatment-related toxicities.

SUMMARY:
This study, called PERSEVERE, examines how local treatment for early breast cancer affects people's health and daily lives over time.

People who join the study will have early-stage breast cancer and receive treatment such as surgery and other therapies that are used before or after surgery. The study does not include people with late-stage (metastatic) breast cancer.

Researchers want to learn about short- and long-term side effects that can happen during or after treatment. These may include tiredness, trouble sleeping, emotional distress, pain, or changes in heart or lung function. The study also looks at how these effects impact participants' quality of life.

Participants will be asked to complete surveys about how they feel. They will also have health checks, such as heart tests, lung function tests, and blood samples. Tissue samples from surgery will also be collected.

The goal is to understand better how different people respond to breast cancer treatment and find ways to support long-term recovery.

DETAILED DESCRIPTION:
PERSEVERE is a prospective, multi-modal cohort study designed to evaluate treatment-related toxicities and quality of life in people with stage I-III early breast cancer receiving local therapy in China. Participants will be eligible if they either:

Receive neoadjuvant therapy (such as chemotherapy or targeted therapy) prior to surgery, or

Undergo surgery followed by postoperative adjuvant therapy, including chemotherapy, radiotherapy, endocrine therapy, or targeted therapy.

The study does not include individuals with recurrent or metastatic breast cancer.

Study Objectives and Methods This study aims to understand the short- and long-term physical, psychological, and social effects of breast cancer treatment and how they impact participants' recovery and daily life.

At baseline, the study collects comprehensive information on participants':

Sociodemographic status: marital status, education level, and household income

Anthropometric measurements: height, weight, body mass index (BMI), waist and hip circumference

Medical history: personal medical history, comorbidities, and past treatments

Reproductive history: menstrual and fertility history

Participants also undergo baseline clinical assessments, including:

Echocardiography (e.g., LVEF) to screen for cardiotoxicity

Pulmonary function testing, conducted for participants aged 70 or older

Routine laboratory tests, such as liver and kidney function, lipid metabolism, and inflammation markers

Biospecimens collected at baseline include:

Peripheral blood (plasma and PBMCs)

Tumor and adjacent normal tissue from surgery

These samples are stored for future biomarker discovery, multi-omics analyses, and translational research on treatment-related toxicities.

Following baseline assessments, participants complete a series of validated patient-reported outcome (PRO) questionnaires, which provide insight into their physical symptoms, emotional well-being, and quality of life. These include:

EORTC QLQ-C30 and QLQ-BR23 for cancer-related quality of life

HADS (Hospital Anxiety and Depression Scale)

Pittsburgh Sleep Quality Index (PSQI) for sleep disturbances

Brief Pain Inventory - Short Form (BPI-SF)

Perceived Stress Scale (PSS-10) for psychological stress

Social Support Rating Scale (SSRS) for social support assessment

Follow-up and Data Collection

Participants are followed using standardized electronic questionnaires administered via the REDCap platform at:

Postoperative week 1, month 1, month 3, and every 6-12 months thereafter for up to 5 years

No repeat biospecimen or clinical tests are collected after baseline. Follow-up focuses on tracking changes in symptoms and quality of life through PROs, enabling analysis of individual recovery trajectories.

Quality Assurance Data collection uses REDCap with built-in logic and range validation

A structured data dictionary ensures consistency across sites

SOPs guide recruitment, consent, biospecimen handling, adverse event reporting, and data entry

Source data verification will be conducted on a sample of participants

Missing data will be managed using statistical imputation and sensitivity analysis

Study Innovation and Impact

PERSEVERE is one of the first large-scale prospective cohort studies in China specifically focused on treatment-related toxicities and quality of life in breast cancer patients. It is designed to:

Capture a comprehensive picture of treatment-related toxicities, beyond acute effects

Enable integrative analysis of biological, physical, and psychological indicators

Build a clinical-biological dataset for developing prediction tools and AI-driven recovery models

Guide personalized supportive care strategies based on Chinese breast cancer patients' needs

The findings will provide new insights into survivorship and recovery and help clinicians deliver evidence-based, patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Diagnosed with stage I, II, or III invasive breast cancer confirmed by pathology or cytology
* No signs of metastatic disease (cancer that has spread to other parts of the body)
* Scheduled to receive local treatment, including:

Surgery

And/or neoadjuvant or adjuvant therapy such as chemotherapy, radiation, hormone therapy, or targeted therapy

* Willing and able to complete health questionnaires and attend follow-up visits
* Has given written informed consent to join the study

Exclusion Criteria:

* Have metastatic breast cancer or local recurrence
* Have already received curative treatment (surgery, chemo, etc.) for the current breast cancer before joining the study
* Are currently pregnant or breastfeeding
* Have a history of another cancer within the past 5 years (except for non-melanoma skin cancer or in-situ cervical cancer)
* Are unable to participate in the study due to mental, physical, or legal reasons (for example, under legal guardianship or imprisonment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from multiple hospitals across China. The study is coordinated by the Cancer Hospital, Chinese Academy of Medical Sciences (CAMS), and includes collaborating sites such as Shanxi Cancer Hospital and the CAMS Cancer Hospital Shenzhen branch. Additional centers from both northern and southern regions of China will be added as the study expands. The study population includes women diagnosed with stage I-III breast cancer who are receiving local therapy in real-world clinical settings across diverse geographic areas.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline, 1week, 1 month, 3 months, 6 months, 12 months, annually up to 5 years
  Quality of life will be measured using the EORTC QLQ-C30, a 30-item questionnaire that includes a global health status/QoL scale, five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, nausea/vomiting, pain), and several single-item symptom measures.
  Score range: Each scale is transformed to a 0-100 scale.
  Interpretation: For functional and global health status scales, higher scores indicate better functioning or quality of life. For symptom scales, higher scores indicate worse symptom burden.
  Changes from baseline will be analyzed across follow-up timepoints.

SECONDARY OUTCOMES:
Trajectories and Risk Factors for Cancer-Related Fatigue Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Fatigue Module (EORTC QLQ-FA12) | Baseline, 1 week, 1 month, 3 months, 6 months, 12 months, then annually up to 5 years
  Cancer-related fatigue will be assessed using the EORTC QLQ-FA12, a 12-item validated module measuring fatigue in three dimensions: physical, emotional, and cognitive.
  Score range: Each dimension is linearly transformed to a score from 0 to 100.
  Interpretation: Higher scores indicate greater fatigue (worse outcome). This outcome will track changes in fatigue over time and examine associations with clinical, biological, and psychosocial factors.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Fang, MD, Principal Investigator — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing 100021, China.
Locations (3):
- China (3):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
PERSEVERE will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: We will consider access to study data upon written detailed request sent to us, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from the study for personal access, and data will only be transferred after signing of a data access agreement.